CLINICAL TRIAL: NCT05933096
Title: Contrast-enhanced Multispectral Optoacoustic Tomography for Functional Assessment of the Gastrointestinal Transit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Ferdinand Knieling, Dr. med. habil Ferdinand Knieling, University of Erlangen-Nürnberg Medical School
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 23-247-Bm
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Gastrointestinal Motility

STUDY DESIGN:
Intervention Model Description: Subjects will ingest three different standardized meals called breakfast 1, breakfast 2, and breakfast 3. They will ingest one meal per day, there is a minimum of 48 hours between measurement days. Every subject will ingest every meal.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Breakfast 1 (Experimental): Breakfast 1 is composed of 500 ml of water, mixed with 50 mg of ICG
  Interventions: Diagnostic Test: Contrast-enhanced multispectral optoacoustic tomography
- Breakfast 2 (Experimental): Breakfast 2 is composed of 200ml of yoghurt, mixed with 50 mg of ICG
  Interventions: Diagnostic Test: Contrast-enhanced multispectral optoacoustic tomography
- Breakfast 3 (Experimental): Breakfast 3 is composed of two slices white toast, two fried eggs and 30 g of jam, mixed with 50 mg of ICG
  Interventions: Diagnostic Test: Contrast-enhanced multispectral optoacoustic tomography

INTERVENTIONS:
Diagnostic Test: Contrast-enhanced multispectral optoacoustic tomography — Ingestion of ICG-labeled food and 10 measurements with MSOT, 1 before ingestion of food, 8 afterwards, each after 60 minutes, 1 measurement 24 hours after ingestion

SUMMARY:
This clinical trial aims to characterize a novel method of imaging the gastrointestinal tract in healthy subjects. The method is using laser-light and soundwaves and it is performed in a similar manner as conventional ultrasound. It is radiation-free and non-invasive.

Participants will ingest food mixed with the clinically-registered dye Indocyanine green. Researchers will measure the signal of the dye over different segments of the gastrointestinal tract, visualizing gastrointestinal transit.

DETAILED DESCRIPTION:
This clinical trial aims to assess gastrointestinal transit by using contrast-enhanced multispectral optoacoustic tomography (MSOT). MSOT is able to visualize not only endogenous chromophores like hemoglobin but also exogenous chromophores such as Indocyanine green (ICG). Healthy subjects will ingest three different standardized meals, all of which are mixed with ICG. By measuring the signal intensity of ICG during gastrointestinal transit, gut motility can be assessed non-invasive and radiation free.

The goal is to compare transit times for different standardized meals, which are liquid, mushy, and solid.

ELIGIBILITY:
Inclusion criteria

* Age over 18 years
* Written informed consent

Exclusion Criteria:

General:

* Pregnancy
* Breastfeeding mothers
* Tattoo in the area of the examination
* Subcutaneous fat tissue over 3 cm
* Chronic or acute diseases of the gastrointestinal tract or symptoms suggesting such a disease
* Acute diseases requiring treatment
* Lack of written consent

ICG related:

* Known hypersensitivity to ICG, sodium iodide or iodine.
* Hyperthyroidism, focal or diffuse thyroid autonomy.
* Timely close treatment to check thyroid function with ingestion of radioactive iodine (within two weeks before or after the study)
* Impaired renal function
* Taking the following medications: Beta blockers, anticonvulsants, cyclopropane, bisulfite compounds, haloperidol, heroin, meperidine, metamizole, methadone, morphine, nitrofurantoin, opium alkaloids, phenobarbital, phenylbutazone, probenecid, rifamycin, any injection containing sodium bisulfite

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-24 (Estimated)

PRIMARY OUTCOMES:
Transit-times of different segments of the gastrointestinal tract | 2 days
  Transit-times of the gastrointestinal passage

SECONDARY OUTCOMES:
Signal-intensity of ICG | 2 days
  Measured with MSOT in arbitrary units

CONTACTS AND LOCATIONS:
Overall Officials: Ferdinand Knieling, MD, Principal Investigator — Kinder- und Jugendklinik Universitätsklinikum Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided